CLINICAL TRIAL: NCT02093286
Title: Phase IV, Study of Safety Profile Following Pentabio Vaccination in Indonesian Infants
Brief Title: Safety Profile Following Pentabio Vaccination in Indonesian Infants
Status: Completed | Type: Observational
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Other Study IDs: PMS Penta 0414
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Pentabio Vaccine; Safety; Infants; Booster Dose; DTwP/HepB/Hib

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pentabio Vaccine: 1 dose of Pentabio vaccine, 0.5 ml Will be given intramuscularly

SUMMARY:
To assess any serious systemic reaction within 30 minutes after Pentabio immunization

DETAILED DESCRIPTION:
Any local and systemic reaction after Pentabio immunization

ELIGIBILITY:
Inclusion Criteria:

* Immunization with Pentabio vaccine
* Parents already understood the consequences to be involved in this study and having signed the informed consent form
* Parents agree and willing to fill in the Diary Card, to record all the reactions after immunization

Exclusion Criteria:

* Given simultaneously with other vaccines or with the interval less than 1 month with other vaccination except OPV/IPV.

Ages: 2 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 4000 infants, 2-11 months old From 4 provincial health primary center
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Any serious adverse event occurring from inclusion until 30 minutes after the injection | 30 minutes
  local and systemic reaction

SECONDARY OUTCOMES:
Percentage of local and systemic events occurring within 72 hours after each injection | 72 hours
  any local and systemics events
Percentage of local and systemic events occurring from 72 hours up to 28 days following injection. | 25 days
  any local and systemic events
Percentage of serious adverse events within 28 days after injection | 28 days
  Any serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Julitasari Sundoro, MD, Principal Investigator — AEFI National Committee
Locations (4):
- Indonesia (4):
  - West Java Provincial Ministry of Health, Bandung, West Java
  - West Nusa Tenggara Provincial Ministry of Health, Mataram, West Nusa Tenggara
  - Bali Provincial Ministry of Health, Bali
  - Yogyakarta Provincial Ministry of Health, Yogyakarta